CLINICAL TRIAL: NCT03139526
Title: Social Participation After Childhood Craniopharyngioma
Acronym: CRANIO
Status: Completed | Type: Observational
Sponsor: BERTHILLIER Julien (Other)
Responsible Party: Sponsor-Investigator, BERTHILLIER Julien, Project Manager, Hospices Civils de Lyon
Organization: Hospices Civils de Lyon (Other)
Other Study IDs: 2015-018
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Children With a Craniopharyngioma
Keywords: Craniopharyngioma; Children; Social participation; Life-H questionnaire
MeSH Terms: conditions — Craniopharyngioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study so no intervention — observational study, so no intervention

SUMMARY:
Craniopharyngioma is a rare, benign central nervous system tumor, which may be a source of multiple complications, from endocrinology to vision, neurology and neurocognitive functions. This morbidity can lead to reduced participation in life activities, as described in the International Classification of Functioning, Disability, and Health (ICF). The primary objective of this study is to measure participation in life activities in a population of children affected by childhood craniopharyngioma, using the assessement of life habits questionnaire (LIFE-H questionnaire), validated as a social participation measurement tool in various pediatric disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Children with a craniopharyngioma

Exclusion Criteria:

* None

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients hospitalized in the pediatric neurosurgery department of Hospices Civils de Lyon between 2007 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
LIFE-H questionnaire (Assessment of Life Habits) | At maximum 6 months after inclusion
  The LIFE-H questionnaire is sent by mail to parents' patient. For parents who do not return the questionnaire completed, a telephone call is made and the LIFE-H questionnaire is completed by phone.

IPD SHARING:
Plan to Share IPD: No